CLINICAL TRIAL: NCT04450667
Title: Impact of Preoperative Oral Rehydration on the Incidence of Spinal Anesthesia-induced Hypotension for Scheduled Cesarean Section.
Brief Title: Post Spinal Anesthesia Hypotension and Preoperative Hydration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Denis SCHMARTZ, Head of department, anesthesiology, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHUB_MATHYPOTA
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia, Spinal; Cesarean Section

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting (No Intervention): Patient will be "nil per os" from midnight before their cesarean section
- Rehydration (Active Comparator): Patient will receive 400 mL of Nutricia Preop ® 2 hours before their cesarean section
  Interventions: Dietary Supplement: Nutricia PreOp

INTERVENTIONS:
Dietary Supplement: Nutricia PreOp — Oral rehydration 2 hours before the scheduled cesarean section under spinal anesthesia
  Arms: Rehydration

SUMMARY:
Study of the impact of preoperative oral rehydration on the incidence of spinal anesthesia-induced hypotension for scheduled cesarean section.

DETAILED DESCRIPTION:
What is already known ? Arterial hypotension is one of the most common complications following spinal anesthesia (60%). Several measures have been studied to prevent this hypotension, such as intravenous vascular filling (preloading, coloading), using different filling fluids (colloids vs crystalloids), preventive administration of vasopressors, reduction of doses and volumes administered in spinal anesthesia.

Only one study has evaluated the impact of oral rehydration on hypotension after spinal anesthesia.

Hypothesis:

The investigatord wish to demonstrate that an oral rehydration 2 hours before surgery, reduces by 50% the incidence of hypotension and / or the use of vasopressors, after spinal anesthesia

Primary outcome:

Decrease in the incidence of hypotension and / or use of vasopressor agents by 50% in the "rehydration" group compared to the "fasting" group.

Secondary outcomes:

Reduced incidence of nausea / vomiting side effects, effect on umbilical pH, APGAR score, patient satisfaction

Design:

Interventional clinical study. Monocentric, single-blind, randomized, single-blind, controlled trial with 2 groups of 50 patients.

Inclusion criteria:

Patients ≥ 18 years old Scheduled for a scheduled cesarean, under spinal anesthesia Signature of informed consent Single pregnancy of ≥ 36 weeks 150 cm <height <180 cm 50 kg <weight <100 kg

Exclusion criteria:

Patient's refusal Contraindication to spinal anesthesia Allergy to a product used for anesthesia Age < 18 Known or pregnancy-related hypertension Gestational diabetes with insulin or pre-existing diabetes with insulin Total language barrier without possibility of translation ASA ≥ 3

Purpose of the study:

The purpose of this study is to show that oral rehydration 2 hours before the induction of anesthesia reduces the incidence of spinal anesthesia-induced hypotension.

The primary hypothesis is that the oral intake of 400 ml of clear liquids (in the form of a standardized carbohydrate solution, NutriciaPreop®) would reduce the hypovolemia related to the preoperative fasting period, and thus reduce the risk of hypotension following the installation of the block.

Primary outcome:

Decrease the incidence of maternal hypotension and / or the use of vasoactive agents in the "rehydration" group by 50%. The blood pressure will be measured by pneumatic cuff, on the arm, once per minute from the entrance to the operating room until the umbilical cord is clamped, then once every 5 minutes until the end of the procedure

Secondary outcomes:

Assess the incidence and severity of nausea / vomiting, umbilical pH, APGAR score, patient comfort (using a visual analog scale graduated from 1 to 10, as well as a satisfaction score of 1 at 5)

Study design:

This is a prospective interventional, single-blind, unicentric, randomized controlled study comprising 2 arms of 50 patients.

An "oral rehydration" arm in which patients will receive 400ml NutriciaPreop to drink 2 hours before anesthesia, and an "fasting" arm in which patients will be fasting since midnight the day before the intervention. As part of the study, the NutriciaPreop solution is provided free to patients.

Duration of the study Including 1 patient per working day, the study will last 6 months. We are considering to set the duration of the study at 9 months.

Materials and methods After recruitment at the anesthesia consultation and signing of the consent, the randomization is carried out by a member of the medical team not involved in the planned cesarean section.

Randomization is done by a sealed, opaque envelope containing the group and the instructions which will be sent to the midwives of the patient's hospital unit.

"Rehydration" arm: 2 boxes of 200 ml Nutricia PreOp to drink 2 hours before anesthesia "Fasting" arm: patient fasting since midnight the day before the intervention Identical premedication in the 2 groups: metoclopramide 10mg + ranitidine 50 mg in 50 ml of 0.9% NaCl IV, as well as 30 ml of sodium citrate per os, on call in the operating room.

Patients will be equipped with 18G venous catheters with obturators to avoid receiving any maintenance fluid before anesthesia (except premedication) Upon arrival in the operating room, the team performs the usual safety checklist.

Patient monitoring with ECG scope, PNI cuff, Sp02 The anesthesiologist performs the standardized spinal anesthesia: 2.2 ml of hyperbaric bupivacaine 0.5% + 0.5 ml of sufentanil concentration 5 micrograms / ml + 100 microgram of morphine (0.1 ml), for a total volume of 2.8 ml, injected in 30-60 seconds, after reflux of CSF into the L3 / L4 space, previously identified by ultrasound.

At the start of the injection, the anesthesiologist's assistant loads the venous catheter with a coloading of 10 ml / kg (ideal weight) of a Hartmann solution (crystalloid balance containing lactate), then maintenance of 1 ml / kg / h until the umbilical cord is clamped.

For the spinal anesthesia, the patient is placed in a seated position, legs hanging. After this has been done, patient is placed in supine position, except for those with a body mass index greater than 35 kG / m2, which are placed in the "beach chair" position. Patients with a BMI≥35 are installed on a "troop elevation pillow". In all cases a tilt of 10 ° to the left will be applied.

Blood pressure measurement per minute on the cuff. Sensory motor block is tested at 5 and 10 min with cold test (ether) and Pricktest. Finally, the surgeon tests before cutting with a pair of pliers, on the incision area.

Hypotension is defined by a fall of at least 20% in systolic BP compared to the reference systolic BP and / or the need to use a vasoactive drug.

Correction of any decrease in systolic BP by boli of 6 micrograms of Noradrenaline in IVD. Possibility of using another vasoactive drug depending on the clinical situation (choice of responsible anesthesiologist) The analysis will be performed until the umbilical cord is clamped, then, the anesthesiologist wiil follow the standard cesarean management protocol.

The umbilical pH as well as the APGAR score of the newborn will be noted. The patient's nausea / vomiting episodes will also be scored and graded on a scale of 0 to 3 with 0 = no nausea-vomiting, 1: moderate nausea not requiring treatment, 2: moderate nausea responding to treatment, 3: nausea not responding to treatment or vomiting.

A digital scale for assessing patient satisfaction and well-being will be used once preoperatively, after signing the consent, and once postoperatively.

Randomization:

Bloc randomization by bloc of 4.

Statistical analysis:

Based on our incidence of 60% of hypotension, a power analysis shows that 42 patients will be needed in each group in order de detect a 50% decrease in the incidence of hypotension; with a power of 80% and alpha fixed at 0.05. 8 patients will be added to each group to compensate for possible dropouts.

Analysis will be done as "intention to treat". Incidence of hypotension will be analyzed by a Chi-square test and the confidence interval will be reported. Secondary outcomes will be analysed by Chi-square test or Fisher's exact test for discontinuous variable and t-test or Mann-Whitney-U test for continuous variables.

A P value < 0.05 will be considered as significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old
* Scheduled for a scheduled cesarean, under spinal anesthesia (CSE)
* Signature of informed consent
* Single pregnancy of ≥ 36 weeks
* 150 cm <height <180 cm
* 50 kg <weight <100 kg

Exclusion Criteria:

* Patient's refusal
* Contraindication to spinal anesthesia
* Allergy to a product used for anesthesia
* Age < 18
* Known or pregnancy-related hypertension
* Gestational diabetes with insulin or pre-existing diabetes with insulin
* Total language barrier without possibility of translation
* ASA ≥ 3

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Hypotension reduction | 60 minutes
  We aim for a 50% reduction in the incidence of hypotension following spinal anesthesia for scheduled C-section.

SECONDARY OUTCOMES:
N+/V+ | 60 minutes
  Incidence of nausea and/or vomiting
Umbilical pH | 60 minutes
  Umbilical pH

OTHER OUTCOMES:
Patients' satisfaction | 24 hours
  Patients' satisfaction measured by a questionary

CONTACTS AND LOCATIONS:
Overall Officials: Denis Schmartz, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Havas F, Orhan Sungur M, Yenigun Y, Karadeniz M, Kilic M, Ozkan Seyhan T. Spinal anesthesia for elective cesarean section is associated with shorter hospital stay compared to general anesthesia. Agri. 2013;25(2):55-63. doi: 10.5505/agri.2013.42204. PMID 23720079
- [Background] American Society of Anesthesiologists Committee. Practice guidelines for preoperative fasting and the use of pharmacologic agents to reduce the risk of pulmonary aspiration: application to healthy patients undergoing elective procedures: an updated report by the American Society of Anesthesiologists Committee on Standards and Practice Parameters. Anesthesiology. 2011 Mar;114(3):495-511. doi: 10.1097/ALN.0b013e3181fcbfd9. No abstract available. PMID 21307770
- [Background] Itoh S, Arai M, Kuroiwa M, Ando H, Okamoto H. [Effect of Preoperative Oral Rehydration on the Hypotension during Spinal Anesthesia.]. Masui. 2016 Sep;65(8):786-789. Japanese. PMID 30351587
- [Background] Awad S, Varadhan KK, Ljungqvist O, Lobo DN. A meta-analysis of randomised controlled trials on preoperative oral carbohydrate treatment in elective surgery. Clin Nutr. 2013 Feb;32(1):34-44. doi: 10.1016/j.clnu.2012.10.011. Epub 2012 Nov 7. PMID 23200124
- [Background] Banerjee A, Stocche RM, Angle P, Halpern SH. Preload or coload for spinal anesthesia for elective Cesarean delivery: a meta-analysis. Can J Anaesth. 2010 Jan;57(1):24-31. doi: 10.1007/s12630-009-9206-7. Epub 2009 Oct 27. PMID 19859776
- [Background] Kim J, Adhikari M, Dhamane S, Hagstrom AE, Kourentzi K, Strych U, Willson RC, Conrad JC. Detection of viruses by counting single fluorescent genetically biotinylated reporter immunophage using a lateral flow assay. ACS Appl Mater Interfaces. 2015 Feb 4;7(4):2891-8. doi: 10.1021/am5082556. Epub 2015 Jan 23. PMID 25581289